CLINICAL TRIAL: NCT02141711
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Sequential-Panel, Multiple Repeat Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAK-438 in Healthy Non-Japanese Male Subjects
Brief Title: TAK-438 - Safety, Blood Levels & Effects of Repeated Doses
Acronym: TAK-438_107
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: TAK-438_107; U1111-1153-8443 (Other: World Health Organization); 2008-004975-22 (EudraCT Number); NCT01873209 (obsolete NCT alias)
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Erosive Esophagitis(EE); Gastroesophageal Reflux Disease (GERD)
Keywords: Drug therapy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1: TAK-438 10 mg (Experimental): TAK-438 10 mg tablets, orally, once, daily, for 7 days.
  Interventions: Drug: TAK-438
- Cohort 2: TAK-438 20 mg (Experimental): TAK-438 20 mg tablets, orally, once, daily, for 7 days.
  Interventions: Drug: TAK-438
- Cohort 3: TAK-438 40 mg (Experimental): TAK-438 40 mg tablets, orally, once, daily, for 7 days.
  Interventions: Drug: TAK-438
- Cohort 4: TAK-438 30 mg (Experimental): TAK-438 30 mg tablets, orally, once, daily, for 7 days.
  Interventions: Drug: TAK-438
- Cohorts 1-4: Placebo (Placebo Comparator): TAK-438 placebo-matching tablets, orally, once, daily, for 7 days.
  Interventions: Drug: TAK-438 Placebo

INTERVENTIONS:
Drug: TAK-438 — TAK-438 tablets
  Arms: Cohort 1: TAK-438 10 mg; Cohort 2: TAK-438 20 mg; Cohort 3: TAK-438 40 mg; Cohort 4: TAK-438 30 mg
Drug: TAK-438 Placebo — TAK-438 placebo-matching tablets
  Arms: Cohorts 1-4: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of TAK-438 in healthy, non-Japanese men male subjects following a randomized, double blind, placebo controlled, sequential panel, multiple-dose schedule.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-438. TAK-438 is being tested to find a safe and well-tolerated dose. This study looked at pharmacokinetic (effect of the body on the drug) and pharmacodynamic properties (effect of the drug on the body) as well as look at lab results and side effects in people who took TAK-438. This study was designed as a randomized, sequential-panel, multiple repeat dose study.

The study population consisted of 4 Cohorts with 12 participants in each Cohort; with 9 participants randomized to receive a single dose of TAK-438, and 3 participants to receive placebo. Participants in each Cohort received a single dose of study drug once daily after a 10-hour fast. The starting dose was 10 mg followed by administrations of 20, 40, and 30 mg.

This single-centre trial was conducted in the United Kingdom. The overall time to participate in this study was up to 37 days. Participants made 2 visits to the clinic for screening, one 11-day period of confinement to the clinic, and 2 further visits after the confinement period. All participants were contacted by telephone 7 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18 to 45, inclusive, who are in good health, as determined by medical history, physical examination, clinical laboratory evaluations and urine drug screen.
* The subject has the ability to tolerate the pH probe for 24 hours prior to Randomization (Day 1).

Exclusion Criteria:

* Clinically significant history of hypersensitivity to any drug or food or any excipients of TAK-438
* History of gastroesophageal reflux disease (GERD), symptomatic GERD, erosive esophagitis, duodenal ulcer,gastric ulcer, dyspepsia, Barrett's esophagus, or Zollinger-Ellison syndrome
* The subject has a positive test result for Helicobacter pylori at the Initial Screening Visit
* Any clinically significant results from physical examinations or clinical laboratory results as deemed by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Days 1 and 7
  (AUC(0-tlqc) is a measure of total plasma exposure to the drug from time 0 to time of the last quantifiable concentration (AUC[0-tlqc]).
AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Days 1 and 7
  AUC(0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
AUC(0-tau): Area Under the Plasma Concentration-time Curve from Time 0 to Time tau Over the Dosing Interval for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Days 1 and 7
  AUC(0-tau) is a measure of the area under the plasma concentration-time curve from time 0 to time tau over a dosing interval, where tau is the length of the dosing interval.
Cmax: Maximum Observed Plasma Concentration for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Days 1 and 7
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Cmin,ss: Minimum Observed Plasma Concentration at Steady State for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Day 7
Cmax,ss: Maximum Observed Plasma Concentration at Steady State for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Day 7
(Cmax-Cmin)/Cavg: Fluctuation of Concentration at Steady State for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Day 7
  (Cmax-Cmin)/Cavg, where Cmin is the minimum observed plasma concentration and Cavg is the average plasma concentration at steady state.
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Days 1 and 7
  Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Terminal Elimination Rate Constant (λz) for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Days 1 and 7
  Terminal elimination rate constant (λz) is the rate at which drugs are eliminated from the body.
Terminal Elimination Half-life (T1/2) Pharmacokinetic Parameter for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Days 1 and 7
  Terminal Phase Elimination Half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Apparent Clearance (CL/F) Pharmacokinetic Parameter for TAK-438 | Days 1 and 7
  CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided AUC(0-24), expressed in L/hr.
Apparent Volume of Distribution (Vz/F) for TAK-438 | Days 1 and 7
  Vz/F is the distribution of a drug between plasma and the rest of the body following oral administration, calculated as CL/F divided by λz.
Ae(0-t): Total Amount of Drug Excreted in Urine from Time 0 to Time T for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Day 1 and Day 7
  Ae(0-t) is the total amount of drug excreted in urine from time 0 to t, where t is 24 hours on Day 1 and 48 hours on Day 7.
Ae(0-tau): Total Amount of Drug Excreted in Urine from Time 0 to Time tau for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Day 1 and Day 7
  Ae(0-tau) is the total amount of drug excreted in urine from time 0 to tau, where tau equals 24 hours.
Renal Clearance (CLr) for TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul | Day 1 and Day 7
  CLr is a measure of apparent clearance of the drug from the urine calculated as total amount excreted in the urine from time 0 to 24 hours postdose / plasma area under the curve from time 0 to 24 hours post-dose.
Fraction of TAK-438 and TAK-438 metabolites M-I, M-II, M-III and M-IV-Sul Excreted in Urine (Fe) | Day 1 and Day 7
  Fe is a measure of the fraction of drug excreted in urine and is calculated as Fe = (total amount excreted in the urine from time 0 to 24 hours post-dose / dose)×100.
Physical Examination Findings | Baseline up to Day 9
  A baseline physical examination (defined as the pretreatment assessment immediately prior to the start of study drug) will consist of the following body systems: (1) eyes; (2) ears, nose, throat; (3) cardiovascular system; (4) respiratory system; (5) gastrointestinal system; (6) dermatologic system; (7) extremities; (8) musculoskeletal system; (9) nervous system; (10) lymph nodes; (11) genitourinary system; and (12) other. All subsequent physical examinations should assess clinically significant changes from the baseline examination.
Number of Participants With Potentially Clinically Significant Vital Sign Findings | Baseline up to Day 9
  Participants with at least one potentially clinically significant post-baseline vital sign finding. Vital signs will include body temperature (oral temperature), sitting blood pressure (after sitting for 5 minutes), and pulse (bpm).
Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings | Baseline to Day 9
  Full 12-lead ECGs will be recorded using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (using Bazett correction; QTcB) intervals. The investigator or other qualified physician will interpret each ECG using one of the following categories: within normal limits, abnormal but not clinically significant, or abnormal and clinically significant.
Number of Participants With Potentially Clinically Significant Laboratory Evaluation Findings | Baseline up to Day 9
  Laboratory tests for hematology, serum chemistries, coagulation tests, and urinalysis will be performed.
Number of Participants With Treatment-Emergent Adverse Events (AEs) | Baseline up to Day 9
  Treatment-emergent adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 7 days after the last dose of study drug, or if a serious adverse event, within 30 days after the last dose of study drug.
Safety of TAK-438 | 3 months
  Assessed by physical examination, ECG, and safety tests of blood/urine
Tolerability of TAK-438 | 3 months
  Assessed by adverse events
Pharmacokinetic analysis of plasma TAK-438 concentrations | 3 months
  Primary pharmacokinetic parameters (AUC (0-tlqc), AUC (0-inf), Cmax) for TAK-438 and its metabolites M-I, M-II, M-III and M-IV-Sul will be subject to statistical analysis
Pharmacodynamic measurement for assay of gastric pH, measurement of gastrin, pepsinogen I, pepsinogen II and the pepsinogen I/II ratio in plasma samples | 3 months

SECONDARY OUTCOMES:
Percentage of Time the pH is Greater than pH 4 and pH 5 over a 24 Hour Period | Over a 24-hour period at Baseline and over a 24-hour period following the administration of study on Days 1, 4 and 7
  Using a calibrated gastric pH monitor, the measurement of stomach pH will be made continuously over a 24-hour period at Baseline and over a 24-hour period following the administration of study on Days 1, 4 and 7.
Percentage of Time the pH is Greater than pH 4 and pH 5 over a 48 Hour Period | Over a 48-hour period following the administration of study on Day 7
  Using a calibrated gastric pH monitor, the measurement of stomach pH will be made continuously over a 48-hour period following the administration of study drug on Day 7.
Percentage of Time the PH is Greater than pH 4 and pH 5 from 8 PM to 8 AM | Over a 12-hour period from 8 PM to 8 AM on Days 1, 4 and 7
  Using a calibrated gastric pH monitor, the measurement of stomach pH will be made continuously over a 12-hour period from 8 PM to 8 AM to assess nocturnal pH.
Total Amount of Gastrin in Plasma | Predose Days 1 through 7 and Days 8 and 9
Total Amount of Pepsinogen I in Plasma | Predose Days 1 through 7 and Days 8 and 9
Total Amount of Pepsinogen II in Plasma | Predose Days 1 through 7 and Days 8 and 9
Pepsinogen I/II Ratio in Plasma | Predose Days 1 through 7 and Days 8 and 9

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda; Steve Warrington, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

REFERENCES:
- [Derived] Jenkins H, Sakurai Y, Nishimura A, Okamoto H, Hibberd M, Jenkins R, Yoneyama T, Ashida K, Ogama Y, Warrington S. Randomised clinical trial: safety, tolerability, pharmacokinetics and pharmacodynamics of repeated doses of TAK-438 (vonoprazan), a novel potassium-competitive acid blocker, in healthy male subjects. Aliment Pharmacol Ther. 2015 Apr;41(7):636-48. doi: 10.1111/apt.13121. Epub 2015 Feb 23. PMID 25707624